CLINICAL TRIAL: NCT03731481
Title: Comparing the Effectiveness of Two Virtual Lifestyle Medicine Interventions Across Urban and Rural Settings
Brief Title: Virtual Lifestyle Medicine Comparative Effectiveness Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Live Healthy Appalachia (Unknown); Ardmore Institute of Health (Other); OhioHealth (Other); Lifestyle Medicine Institute (Unknown)
Responsible Party: Principal Investigator, David Drozek, Assistant Professor of Surgery, Heritage College of Osteopathic Medicine, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-X-166
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Chronic Disease; Obesity; Sleep Disorder; Depression
MeSH Terms: conditions — Chronic Disease; Obesity; Sleep Wake Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness research of two interventions across four cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CHIP - Urban (Experimental): Participants randomized by urban location of residence to receive CHIP Lifestyle Medicine program intervention.
  Interventions: Behavioral: Lifestyle Medicine
- CHIP - Rural (Experimental): Participants randomized by rural location of residence to receive CHIP Lifestyle Medicine program intervention.
  Interventions: Behavioral: Lifestyle Medicine
- FPD2- Urban (Experimental): Participants randomized by urban location of residence to receive FPD2 Lifestyle Medicine program intervention.
  Interventions: Behavioral: Lifestyle Medicine
- FPD2 - Rural (Experimental): Participants randomized by rural location of residence to receive FPD2 Lifestyle Medicine program intervention.
  Interventions: Behavioral: Lifestyle Medicine

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle Medicine programs provide instruction in plant-based nutrition, food preparation, methods of stress reduction and incorporation of physical activity into daily routine.

SUMMARY:
This study evaluates the effectiveness of two online Lifestyle Medicine programs. Participants will be randomized by residence, urban vs. rural, into one of two Lifestyle Medicine programs.

DETAILED DESCRIPTION:
This study compares the effectiveness of two virtual Lifestyle Medicine programs across two settings: urban and rural. Program materials include nutritional education, methods to reduce personal stress, and incorporation of physical activity in daily routine. Bio-marker and subjective/self-reported survey measures will be collected at baseline, 5-weeks and six-months from baseline. Study seeks to measure variations in participant outcomes across two lifestyle interventions, participant engagement and level of adherence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to read and write English
* Access to high-speed Internet
* Taking medication for at least one chronic disease condition such as high blood pressure, OR are overweight (BMI of 25 or greater)
* Willing to provide blood samples at three time points
* Willing to complete online surveys at three time points

Exclusion Criteria:

* Advised by physician to limit physical activity
* Previous experience with lifestyle medicine programs, specifically Lifestyle Medicine Clinic, Complete Health Improvement Program, Full Plate Diet
* Household includes someone who has previous experience with a Lifestyle Medicine program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Level of participant engagement | 6 months
  Measure of number of sign-ins and class attendance

SECONDARY OUTCOMES:
Chronic disease status | Baseline, 5-weeks, and 6-months from baseline
  Change in medication dosage for chronic disease conditions
Psychological status | Baseline, 5-weeks, and 6-months from baseline
  Change in psychological state from self-reported, validated surveys

CONTACTS AND LOCATIONS:
Overall Officials: David Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No